CLINICAL TRIAL: NCT00272675
Title: Prevention of Nosocomial Infection in Cardiac Surgery by Decontamination of the Naso- and Oropharynx With Chlorhexidine. A Randomized, Double-Blind, Placebo-Controlled Clinical Trial.
Brief Title: Prevention of Nosocomial Infection by Decontamination of the Naso- and Oropharynx With Chlorhexidine (NONI Trial)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Onze Lieve Vrouwe Gasthuis (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WO-03.021
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2006-01-09 (Estimated); Status verified 2006-01

CONDITIONS: Nosocomial Infection; Respiratory Tract Infection; Surgical Site Infection
Keywords: Nosocomial infection,; Decontamination,; Randomized placebo-controlled trial,; Cardiac surgery,; Chlorhexidine,; Prevention
MeSH Terms: conditions — Cross Infection; Respiratory Tract Infections; Surgical Wound Infection | interventions — chlorhexidine gluconate; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Chlorhexidine gluconate (drug) vs placebo

SUMMARY:
Does chlorhexidine gluonate, a simple broad-spectrum antimicrobial agent with virtually no adverse-effects lower the incidence of NI after cardiac surgery, especially with respect to LTI and SSI?

DETAILED DESCRIPTION:
Nosocomial infections (NIs) after open heart surgery are recognized as an important cause of morbidity and mortality with a prolonged hospital stay, increased need for of antibiotics, decreased quality of life and higher concomitant costs. Decontamination of the oropharynx seems important, since there is direct evidence of an association between pulmonary infection and oral health. Another important strategy involves the eradication of Staphylococcus aureus, the most important pathogen causing SSI. The most common reservoir of S.aureus is the anterior nares and eradication can be achieved by the application of topical antibiotics. Although promising results have been reported for both strategies, they are not widely used as routine prevention methods because of the variability of trial design, the concern about the emergence of antimicrobial resistance and increased costs. Further research is essential to evaluate different protocols, antimicrobial agents and cost-effectiveness.

Fur this purpose, we designed a clinical trial to study wether a simple broad-spectrum antimicrobial agent with virtually no adverse-effects would lower the incidence of NI after cardiac surgery, especially with respect to LTI and SSI.

Comparison(s): Oropharyngeal and nasal decontamination with chlorhexidine compared to placebo in patients after cardiothoracic surgery

ELIGIBILITY:
Inclusion Criteria:

* all adult patients (above 18) who were scheduled to undergo sternotomy for cardiothoracic surgery

Exclusion Criteria:

* emergency procedures, a preoperative infection and/or the use of antibiotics, hypersensitivity to chlorhexidine gluconate (CHX), absence of written informed consent or presence of an alternative prophylactic regimen like selective decontamination of the digestive tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2003-08; Study Completion 2005-09

PRIMARY OUTCOMES:
Nosocomial Infection

SECONDARY OUTCOMES:
Respiratory tract and surgical site infection; S. aureus nasal carriage, nonprophylactic antibiotic use, hospital stay, in-hospital mortality, optimal duration of preoperative trial medication and medication adverse-effects.

CONTACTS AND LOCATIONS:
Overall Officials: Patrique Segers, Drs., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Onze lieve vrouwe gasthuis, Amsterdam, Netherlands

REFERENCES:
- [Derived] Segers P, Speekenbrink RG, Ubbink DT, van Ogtrop ML, de Mol BA. [Prevention of nosocomial infections after cardiac surgery by decontamination of the nasopharynx and oropharynx with chlorhexidine; a prospective, randomised study]. Ned Tijdschr Geneeskd. 2008 Mar 29;152(13):760-7. Dutch. PMID 18461895
- [Derived] Segers P, Speekenbrink RG, Ubbink DT, van Ogtrop ML, de Mol BA. Prevention of nosocomial infection in cardiac surgery by decontamination of the nasopharynx and oropharynx with chlorhexidine gluconate: a randomized controlled trial. JAMA. 2006 Nov 22;296(20):2460-6. doi: 10.1001/jama.296.20.2460. PMID 17119142